CLINICAL TRIAL: NCT05380180
Title: Enhancing Quality of Life for Older Adults With and Without Mild Cognitive Impairment (MCI) Through Social Engagement Over Video Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Wendy Rogers, Khan Professor of Applied Health Sciences, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22212
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Aging; Mild Cognitive Impairment; Aging Well
Keywords: videoconferencing; social engagement; loneliness; social isolation; quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Social Isolation

STUDY DESIGN:
Intervention Model Description: Participants will be screened and assigned to either intervention group or wait-listed group.
Who Masked: Investigator
Masking Description: All primary and secondary outcome assessments completed at Week 4 and Week 8 are blinded. Participants are told ahead of time to not share their group information with the blinded assessor during administration of measures. Supplementary outcome measures require the assessor to know the group assignment, as these measures pertain to their current experience in the intervention. Thus, all supplementary outcome measures are administered at a separate time by an unblinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OneClick Social Engagement Intervention Group (Experimental): Intervention group participants will receive the social engagement OneClick intervention for 8 weeks, and will complete a mid-assessment at week 4, and a post-assessment at week 8.
  Interventions: Other: OneClick Social Engagement Intervention
- OneClick Social Engagement Waitlist Control Group (Other): Waitlist control group participants will receive no intervention for the first 8 weeks and will complete assessments at week 4 and week 8. Following the completion of the 8-week controlled portion, waitlist participants will be provided with the opportunity to participate in the OneClick social engagement intervention through the intervention extension.
  Interventions: Other: OneClick Social Engagement Intervention Extension

INTERVENTIONS:
Other: OneClick Social Engagement Intervention — Intervention group participants will receive the social engagement OneClick intervention for 8 weeks, and will complete a mid-assessment at week 4, and a post-assessment at week 8. Participants will use a computer or tablet to participate in two social engagement events per week. The intervention events will be delivered through the OneClick video conferencing platform. During each session participants will watch a short slideshow around a series of topics (e.g., nature, technology, hobbies) and get to engage in conversations surround the topics presented, which will be held in breakout rooms. Breakout room discussions will be set for 30 minutes, and participants will be provided with questions surrounding the topics to help stimulate conversation.
  Arms: OneClick Social Engagement Intervention Group
Other: OneClick Social Engagement Intervention Extension — Waitlist control group participants will receive no intervention for the first 8 weeks and will complete assessments at week 4 and week 8. Following the completion of the 8-week controlled portion, waitlist participants will be provided with the opportunity to participate in the OneClick social engagement intervention through the intervention extension. Waitlist participants will use a computer or tablet to participate in two social engagement events per week. The intervention events will be delivered through the OneClick video conferencing platform over the span of 8 weeks.
  Arms: OneClick Social Engagement Waitlist Control Group

SUMMARY:
The goal of this randomized controlled trial is to rigorously assess the efficacy of an 8-week social engagement OneClick intervention. A total of 120 older adults with and without mild cognitive impairment (60 per group) will be randomized after a baseline assessment to the social engagement OneClick intervention group or the waitlist control group. Participants assigned to the intervention group will receive the social engagement OneClick intervention for 8 weeks, and will complete a mid-assessment at week 4, and a post-assessment at week 8. Participants assigned to the waitlist control group will receive no intervention for the first 8 weeks and will complete assessments at week 4 and week 8. Subsequently, as an extension to this study, participants assigned to the waitlist control group will have an opportunity to participate in 8 weeks of social engagement OneClick intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Fluent in English
* Adequate visual and auditory acuity
* Passing score on Telephone Interview for Cognitive Status - Modified (TICS-M) of 22 and above included
* Passing score on Montreal Cognitive Assessment (MoCA) of 20 and above included
* Geriatric Depression Scale (GDS) score of less than 9
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Access to and ability to use necessary resources for participating in technology-based intervention

Exclusion Criteria:

* Diagnosis of dementia
* Live in assisted living facility or skilled nursing facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A Rogers, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (2):
- United States (2):
  - University of Illinois, Urbana Champaign, Champaign, Illinois
  - CJE Senior Living, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Started | 50 | 49
Completed | 41 | 46
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- OneClick Social Engagement Waitlist Control Group: Waitlist control group participants will receive no intervention for the first 8 weeks and will complete assessments at week 4 and week 8. Following the completion of the 8-week controlled portion, waitlist participants will be provided with the opportunity to participate in the OneClick social engagement intervention through the intervention extension.
  OneClick Social Engagement Intervention Extension: Waitlist control group participants will receive no intervention for the first 8 weeks and will complete assessments at week 4 and week 8. Following the completion of the 8-week controlled portion, waitlist participants will be provided with the opportunity to participate in the OneClick social engagement intervention through the intervention extension. Waitlist participants will use a computer or tablet to participate in two social engagement events per week. The intervention events will be delivered through the OneClick video conferencing platform over the span of 8 weeks. Intervention effects will be measured at week 4 and week 8 of the intervention extension.
- Total: Total of all reporting groups
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (6.3) | 74.6 (7.1) | 74.05 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 46 | 40 | 86
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Isolation Measured by Friendship Scale
Description: Measures six dimensions that contribute to social isolation. Lower scores indicate lower extent of social isolation. Range (0-24)
Time Frame: Baseline, Week 4, Week 8
Population: We implemented an intent-to-treat analysis, including all participants who were randomized in the analysis, regardless of their participation status. To analyze the main effects of the intervention, we conducted linear mixed-effects model. Fixed factors included time of assessment (baseline/Week 4/Week 8) and group (intervention/waitlist control). Participant was included as a random intercept to account for individual variability at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Number analyzed (Participants) | 50 | 49
score on a scale
  Baseline | 20.37 (3.26) | 20.54 (3.30)
  Week 4: number analyzed (Participants) | 41 | 43
  Week 4 | 20.05 (3.31) | 20.23 (3.35)
  Week 8: number analyzed (Participants) | 41 | 46
  Week 8 | 20.39 (3.05) | 19.54 (4.34)
Statistical Analysis 1: Comparison: OneClick Social Engagement Intervention Group vs OneClick Social Engagement Waitlist Control Group; We implemented an intent-to-treat analysis, including all participants who were randomized in the analysis, regardless of their participation status. To analyze the main effects of the intervention, we conducted linear mixed-effects model. Fixed factors included time of assessment (baseline/Week 4/Week 8) and group (intervention/waitlist control). Participant was included as a random intercept to account for individual variability at baseline; Test type: Superiority; p < .05, Mixed Models Analysis

2. Primary Outcome: Change in Loneliness Measured by University of California - Los Angeles (UCLA) Loneliness Scale
Description: Measures the respondents' subjective feeling of loneliness. Higher scores indicate a greater feeling of loneliness. Range (20-80).
Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Number analyzed (Participants) | 50 | 49
score on a scale
  Baseline | 37.93 (8.94) | 37.08 (9.35)
  Week 4: number analyzed (Participants) | 41 | 43
  Week 4 | 40.34 (8.88) | 38.60 (9.35)
  Week 8: number analyzed (Participants) | 41 | 46
  Week 8 | 38.05 (8.92) | 39.00 (9.62)
Statistical Analysis 1: Comparison: OneClick Social Engagement Intervention Group vs OneClick Social Engagement Waitlist Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Mixed Models Analysis

3. Primary Outcome: Change in Quality of Life Measured by Quality of Life in Alzheimer's Disease
Description: Measures quality of life indicators such as physical health, energy, family, and money. Lower scores indicate a lower quality of life. Range (13-52).
Time Frame: Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Number analyzed (Participants) | 50 | 49
score on a scale
  Baseline | 37.52 (5.21) | 37.81 (5.11)
  Week 4: number analyzed (Participants) | 41 | 43
  Week 4 | 36.88 (5.56) | 36.63 (5.52)
  Week 8: number analyzed (Participants) | 41 | 46
  Week 8 | 37.44 (5.48) | 36.54 (5.57)
Statistical Analysis 1: Comparison: OneClick Social Engagement Intervention Group vs OneClick Social Engagement Waitlist Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Mixed Models Analysis

4. Secondary Outcome: Change in Social Network Measured by Lubben Social Network Index
Description: Measures social network size for both family and friends and also the frequency of interaction with them. Higher scores indicate higher level of social engagement. Range (0-30).
Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Number analyzed (Participants) | 50 | 49
score on a scale
  Baseline | 18.75 (4.43) | 19.08 (4.55)
  Week 4: number analyzed (Participants) | 41 | 43
  Week 4 | 17.59 (5.50) | 17.28 (4.90)
  Week 8: number analyzed (Participants) | 41 | 46
  Week 8 | 17.51 (4.50) | 17.54 (4.74)
Statistical Analysis 1: Comparison: OneClick Social Engagement Intervention Group vs OneClick Social Engagement Waitlist Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Mixed Models Analysis

5. Secondary Outcome: Change in Social Activity Measured by Social Activity Frequency
Description: Measures how often during the past year participants have engaged in various social activities. Lower scores indicate less engagement in social activities. Range (10-50).
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
Number analyzed (Participants) | 50 | 49
score on a scale
  Baseline | 26.84 (4.01) | 27.98 (3.98)
  Week 4: number analyzed (Participants) | 41 | 43
  Week 4 | 27.63 (4.08) | 27.89 (5.05)
  Week 8: number analyzed (Participants) | 41 | 46
  Week 8 | 28.07 (4.69) | 27.30 (4.44)
Statistical Analysis 1: Comparison: OneClick Social Engagement Intervention Group vs OneClick Social Engagement Waitlist Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .05, Mixed Models Analysis

6. Other Pre Specified Outcome: Change in System Usability Measured by System Usability Scale
Description: Measures the respondents' perception of usability of the OneClick system. Higher scores indicate higher ease of use and usefulness, and lower scores indicate more difficulty to use the system and decreased usefulness. Range (0-100).
Time Frame: Week 4 of intervention, Week 8 of intervention
Measure: Mean (Standard Deviation); unit: Raw Score
Arm/Group | OneClick Social Engagement Intervention Group
Number analyzed (Participants) | 39
Raw Score
  Change Score at Week 4 | 63.80 (18.7)
  Change Score at Week 8 | 68.20 (18.6)

7. Other Pre Specified Outcome: Change in Technology Acceptance Measured by Technology Acceptance Survey
Description: Measure of technology acceptance: perceived ease of use. Lower scores indicate lower perception of ease of use. Range (1-7).
Time Frame: Week 4 of intervention, Week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group
Number analyzed (Participants) | 39
score on a scale
  Change Score at Week 4 | 5.40 (1.4)
  Change Score at Week 8 | 5.70 (1.2)

8. Other Pre Specified Outcome: Change in Computer Proficiency Measure by Computer Proficiency Questionnaire (Short -Form)
Description: Measures the ability to perform a number of tasks using a computer. Tasks include computer basics, printing, communication, internet, scheduling, and multimedia. Higher scores indicated higher rates of proficiency. Range (6-30).
Time Frame: Week 4 of intervention, Week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OneClick Social Engagement Intervention Group
Number analyzed (Participants) | 39
score on a scale
  Change Score at Week 4 | 27.60 (2.8)
  Change Score at Week 8 | 28.10 (2.6)

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Description: 0
Arm/Group | OneClick Social Engagement Intervention Group | OneClick Social Engagement Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT05380180/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT05380180/SAP_001.pdf